CLINICAL TRIAL: NCT01197053
Title: ARACHILD: A Multicentric, Double Blind Placebo-controlled Pilot Protocol to Study the Efficacy and Safety of an Epicutaneous Immunotherapy in Children Allergic to Peanut
Brief Title: Epicutaneous Immunotherapy in Peanut Allergy in Children
Acronym: ARACHILD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: DBV Technologies (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: P091102; 2010-019541-26 (EudraCT Number); A100293-36 (Other: AFSSAPS)
Record Dates: First submitted 2010-09-07; First posted 2010-09-09 (Estimated); Last update posted 2015-10-20 (Estimated); Status verified 2015-10

CONDITIONS: Peanut Allergy
Keywords: Peanut Allergy; Food Allergy; Epicutaneous Immunotherapy (EPIT); Food Challenge
MeSH Terms: conditions — Peanut Hypersensitivity; Food Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 100 mcg DBV712 (active) (Experimental): 100 mcg DBV712 administered epicutaneously every 24 hours.
  Interventions: Biological: Epicutaneous Immunotherapy
- Placebo (Placebo Comparator): Placebo will be administered epicutaneously every 24 hours
  Interventions: Biological: placebo of peanut

INTERVENTIONS:
Biological: Epicutaneous Immunotherapy — 100 mcg peanut proteins (active arm) applied on the skin every 24 hrs for 6 months blinded, followed by 12 months open treatment for all patients in the active arm
  Arms: 100 mcg DBV712 (active)
Biological: placebo of peanut — placebo applied on the skin every 24 hrs for 6 months blinded, followed by 12 months open treatment for all patients in the active arm
  Arms: Placebo

SUMMARY:
This study aims at showing that Epicutaneous Immunotherapy with peanut proteins is safe and efficacious for desensitizing children with peanut allergy.

DETAILED DESCRIPTION:
Peanut allergy is a common allergy in the United Sates, with prevalence in the general population as high as 1%. Peanut allergy starts in childhood, its prevalence in children has doubled in the past 5 years, and barely 20% of the allergic children will outgrow this allergy So far, the only treatments available for peanut allergy are avoidance of peanut and injectable epinephrine after the allergic systemic reactions have started. Immunotherapy methods currently available have shown some limitations in their use because of important safety issues. Hence, there is an important unmet medical need for efficient and safe treatment of peanut allergy.

DBV Technologies, is a French biotech company which has developed an Epicutaneous Delivery System, called Viaskin®, a method based on delivering precise quantity of allergens on the upper layers of the skin, i.e. on the epidermis and without any passage in the vascularised dermis. Avoiding contact between the allergens and the bloodstream should confer to epicutaneous immunotherapy (EPIT) a high level of safety as systemic reactions are circumvented.

The goal of this pilot study is to demonstrate that epicutaneous immunotherapy (EPIT) with Viaskin® is safe and efficacious for the desensitization of peanut-allergic children, i.e. increasing the quantity of peanut proteins they can consume symptom-free.

Fifty-two (52) children from 5 to 17 years of age with a confirmed peanut allergy during a baseline double blind placebo-controlled food challenge (DBPCFC) (reacting to a capped value below 250 mg of peanut proteins) will be randomized 1 to 1 and treated either with DBV712, the Viaskin® disk loaded with 100 mcg peanut proteins (active treatment), or with placebo, the Viaskin® disk loaded with a placebo formulation devoid of peanut. Each child will receive one application of one Viaskin® on the skin every day repeatedly for 6 months in a blinded manner, followed by a 12-month open treatment with DBV712 for all of them; placebo children will all cross-over after the first 6 months of treatment to also receive the active treatment.

A DBPCFC to peanut will then be conducted after every 6 months of treatment to assess the efficacy of the treatment. Safety will be assessed during the whole study period.

Skin testing, peanut-specific IgE and IgG4 will occur at selected visits

ELIGIBILITY:
Inclusion Criteria:

* Male or Female between 5 and 17 years of age at enrollment
* An efficient contraceptive method for girls with childbearing potential. Acceptable methods include sexual abstinence, oral, injectable contraceptive methods, intra uterine device.
* Negative pregnancy test for girls with childbearing potential.
* Child with a documented allergy to peanut, i.e. with peanut-specific IgE (>5KU/L, ImmunoCAP method) and/or a positive skin prick test to peanut (wheal diameter ≥ 8mm).
* Child able to consume a cumulated quantity of peanut proteins <250 mg during the baseline DBPCFC.
* Child and his/her legal representative(s) who provide a signed consent form and assent form.
* Child and his/her legal representative(s) whose family and social conditions allow them to understand the protocol and agree to comply in the long term with all study requirements.

Exclusion criteria :

* Child considered too severely allergic to peanut: with a history of severe anaphylaxis to peanut (with hypotension, loss of consciousness, severe bradycardia, respiratory or cardiac arrest requiring an admission to emergency rooms).
* Child with peanut-specific IgE<5 KU/L and whose skin prick test to peanut gave a wheal diameter <8mm).
* Child participating or having participated in a therapeutic study in the last 3 months
* Pregnancy or Breastfeeding
* Child with a generalized eczema
* Child with an immune deficiency
* Diabetic child
* Child allergic to chocolate
* Child or legal representative(s) who did not sign their consent or assent
* Child with no baseline DBPCFC
* Child having reacted to placebo during the baseline DBPCFC
* Child able to consume > 250 mg of cumulated peanut proteins during the baseline DBPCFC
* Child with a respiratory deficiency or with an uncontrolled asthma.
* Child who could not discontinue oral or I.V. antihistamines or oral or I.V. corticosteroids at least the week prior to Visit 1.
* Child with important skin lesions precluding the application of the disks.
* Child not affiliated to social security.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2010-08; Primary Completion 2015-02 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Proportion of patients able to consume >1000 mg of peanut proteins symptom-free | 6 months
  Proportion of patients able to consume >1000 mg of peanut proteins symptom-free during the double blind placebo-controlled food challenges (DBPCFC) to peanut at 6 months, or who have a 10-fold increase in the quantity of peanut proteins consumed as compared to baseline value

SECONDARY OUTCOMES:
Description of the level of Ig | 6 months
  * Level of Peanut-specific IgE at 3 months and 6 months in both groups of treatment.
  * Level of Peanut-specific IgG4 at 3 months and 6 months in both groups of treatment.
  * Evolution of peanut-specific IgE between Day-21 and 12 months and between Day-21 and 18 months for each subject in both groups.
  * Evolution of Peanut-specific IgG4 between Day-21 and 12 months and between Day-21 and 18 months for each subject in both groups.
Proportion of patients able to consume >1000 mg of peanut proteins symptom-free | 12 months
  -Proportion of patients able to consume >1000 mg of peanut proteins symptom-free during the double blind placebo-controlled food challenges (DBPCFC) to peanut at 12 months
Proportion of patients able to consume >1000 mg of peanut proteins symptom-free | 18 months
  -Proportion of patients able to consume >1000 mg of peanut proteins symptom-free during the double blind placebo-controlled food challenges (DBPCFC) to peanut at 18 months
diameter and safety | 3, 6, 12 and 18 months
  * Diameter of the wheal of the Skin Prick tests to peanut at month 3 and month 6 in both groups
  * Diameter of the wheal of the Skin Prick tests to peanut at 12 and 18 months for each subject in both groups
  * Safety and tolerability of the epicutaneous administration of peanut proteins to peanut allergic children at 6, 12 and 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Dupont, MD, PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hopital Necker, Paris, France